CLINICAL TRIAL: NCT01996176
Title: Take a Stand ! - a Cluster Randomized Controlled Intervention Study at Four Office-based Workplaces Aiming to Reduce Occupational Sitting Time
Brief Title: Take a Stand! - an Intervention to Reduce Occupational Sitting Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: TRYG Foundation (Other)
Responsible Party: Principal Investigator, Ida Høgstedt Danquah, Research Assistant, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61110-2071
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary Lifestyle; Sedentary work; Office workers; Work; Workplace intervention; Sitting time
MeSH Terms: conditions — Sedentary Behavior | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention group
  Interventions: Behavioral: Intervention group
- Intervention control (Placebo Comparator): Control group
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — The intervention consists of four components, which as described below:
  1. Information about sedentary behaviour and health: Delivered at the kick-off workshop, in a leaflet and the project website.
  2. Local adaptation: Participants adapt the intervention to their personal and local environment setting individual and common goals. Local ambassadors are chosen and support from the management is emphasised.
  3. Structural changes: Facilities for standing meetings, both formal and informal. Routes for walking meetings should be defined.
  4. Individual support: At the kick-off workshop participants set individual goals. The individual can choose to receive e-mails and text messages (SMS)from the project. The individual receives a post-it block and a postcard to remind them of the project.
  Arms: Intervention group
Behavioral: Control group — The control group receives the intervention after the last follow-up, the exact time will be settled together with each workplace in the control group.
  Arms: Intervention control

SUMMARY:
The purpose of the study is to test an intervention aiming to reduce sitting time during work hours among office workers.

Expectations according to outcome measures: Sitting time reduced by 1 hour pr. day (primary). Number of prolonged periods reduced by 1 pr. day (primary). Number of breaks increased by 3 pr. day (primary). 20 % of participants report a reduction of musculoskeletal pain (secondary). A reduction in waist circumference of 1 cm (secondary). A reduction of 0.5 % in bodyfat (secondary).

DETAILED DESCRIPTION:
Background and aim: Sedentary behaviour has substantial impact on wellbeing and health, e.g. on the risk of cardiovascular disease and premature death. These associations seem to apply as well to people who carry out the recommended 30 minutes of physical activity per day. However, studies indicate that the harmful effects can be reduced through breaking prolonged periods of sitting by intervals of standing or walking.

In total 46 % of Danes are working in occupations which are primarily sedentary and the workplace is thus a relevant setting to intervene against sedentary behaviour.

The aim of the study is to test an intervention towards sitting time among office workers. The intervention will target both total sitting time, breaks from sitting and prolonged periods of sitting.

Design: Cluster-randomized control study led at four different workplaces in Denmark and Greenland. Each workplace should consist of four independent sections (clusters) of about 25 people. Those four sections are randomized to intervention or control. A cluster design is used because the intervention will target the workplace setting as a whole, thus individuals within the same office has to be randomized to the same arm of the intervention.

Participants: 400 adults with sedentary office-based work. Subjects should understand Danish and be without disabilities or diseases affecting their ability to stand or walk.

Intervention: Participating clusters are randomized to

1. Intervention: The intervention consists of four parts: Information, local adaptions, structural changes and individual support.
2. Control: The control group will receive the intervention after the last follow-up (about 3 months later).

Methods: Data on sedentary behaviour is collected objectively using ActiGraph. Waist circumference and body fat percentage is measured. Questionnaire data will be collected on background variables, physical activity level, workplace conditions and well-being.

Data will be collected at baseline, and after 1 and 3 months.

Analysis will be carried out following the intention-to-treat principle comparing the intervention and control group. We will use several outcomes and include baseline values as a covariate (ANCOVA). In addition we will use multilevel models to account for the hierarchical structure of data (workplace, cluster and participant).

Process evaluation will be conducted by the use of qualitative interviews and questionnaire data and concern both adoptions, implementation and sustainability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Workplaces should be:

   * Office-based with sedentary workers
   * Able to include four sections of about equal size (about 25 people) and which could be separated to minimize spill-over effects (e.g. four different addresses, buildings or floors).
   * Have a management willing to collaborate about the project by participating at meetings and at kick-off.
   * Should have at least some financial resources to make structural changes at the work place.
2. Individuals should be:

   * Adults >18 years
   * Sedentary office-based work-
   * Understanding of Danish
   * Without sickness or disabilities affecting their ability to stand or walk
   * Not pregnant
   * Working more than 4 days a week (>30 h)

Exclusion Criteria:

* Not providing signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reduced total time spend sitting at work | 1 month
  Method of measurement: ActiGraph, average daily sitting time during work hours.
Reduced number of prolonged siting periods (>30 min) | 1 month
  Method of measurement: ActiGraph, number of periods sitting >30 min.
Increased number of breaks from sitting time | 1 month
  Method of measurement: ActiGraph, number of postural shifts from sitting to standing/walking

SECONDARY OUTCOMES:
Reduced musculoskeletal problems | 1 month
  Method of measurement: Questionnaire
Waist circumference | 3 month
  Method of measurement: Waist circumference measurement
Body fat percentage | 3 months
  Method of measurement: Body fat % is measured using a segmental body composition analyser
Reduced total time spend sitting at work | 3 months
  Method of measurement: ActiGraph, average daily sitting time during work hours
Reduced number of prolonged siting periods (>30 min) | 3 months
  Method of measurement: ActiGraph, number of periods sitting >30 min
Increased number of breaks from sitting time | 3 months
  Method of measurement: ActiGraph, number of postural shifts from sitting to standing/walking

CONTACTS AND LOCATIONS:
Overall Officials: Janne S Tolstrup, MD, PhD, Study Director — National Institute of Public Helath - University of Southern Denmark; Morten Grønbæk, MD PhD, Study Chair — Centre for Intervention Research in HEalth Promotion and Disease Prevention
Locations (1):
- National Institute of Public Health - University of Southern Denmark, Copenhagen, Denmark

REFERENCES:
- [Result] Danquah IH, Kloster S, Holtermann A, Aadahl M, Bauman A, Ersboll AK, Tolstrup JS. Take a Stand!-a multi-component intervention aimed at reducing sitting time among office workers-a cluster randomized trial. Int J Epidemiol. 2017 Feb 1;46(1):128-140. doi: 10.1093/ije/dyw009. PMID 27094749
- [Derived] Danquah IH, Kloster S, Tolstrup JS. "Oh-oh, the others are standing up... I better do the same". Mixed-method evaluation of the implementation process of 'Take a Stand!' - a cluster randomized controlled trial of a multicomponent intervention to reduce sitting time among office workers. BMC Public Health. 2020 Aug 8;20(1):1209. doi: 10.1186/s12889-020-09226-y. PMID 32770969
- [Derived] Danquah IH, Tolstrup JS. Does It Work for Everyone? The Effect of the Take a Stand! Sitting-Intervention in Subgroups Defined by Socio-Demographic, Health-Related, Work-Related, and Psychosocial Factors. J Occup Environ Med. 2020 Jan;62(1):30-36. doi: 10.1097/JOM.0000000000001737. PMID 31626067
- [Derived] Danquah IH, Pedersen ESL, Petersen CB, Aadahl M, Holtermann A, Tolstrup JS. Estimated impact of replacing sitting with standing at work on indicators of body composition: Cross-sectional and longitudinal findings using isotemporal substitution analysis on data from the Take a Stand! study. PLoS One. 2018 Jun 13;13(6):e0198000. doi: 10.1371/journal.pone.0198000. eCollection 2018. PMID 29897943
- [Derived] Danquah IH, Kloster S, Holtermann A, Aadahl M, Tolstrup JS. Effects on musculoskeletal pain from "Take a Stand!" - a cluster-randomized controlled trial reducing sitting time among office workers. Scand J Work Environ Health. 2017 Jul 1;43(4):350-357. doi: 10.5271/sjweh.3639. Epub 2017 Apr 3. PMID 28368549
- [Derived] Pedersen ES, Danquah IH, Petersen CB, Tolstrup JS. Intra-individual variability in day-to-day and month-to-month measurements of physical activity and sedentary behaviour at work and in leisure-time among Danish adults. BMC Public Health. 2016 Dec 3;16(1):1222. doi: 10.1186/s12889-016-3890-3. PMID 27914468